CLINICAL TRIAL: NCT06236607
Title: Hybrid Closed Loop Effectiveness Trial in Adults With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-44351; 1R01DK138309-01 (NIH)
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Complications
Keywords: Hybrid closed loop (HCL); HCL pump therapy; Multiple daily injections (MDI); Continuous glucose monitoring (CGM); Glucose time-in-range (TIR); Glucose management indicator (GMI); Diabetic ketoacidosis; Patient reported outcomes (PRO); Ecological momentary assessment (EMA)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications; Diabetic Ketoacidosis

STUDY DESIGN:
Intervention Model Description: The trial will have a four-arm, parallel group design, with 9-month intervention phase. Adults with T1D on MDI therapy will be randomized in a 1:1:1:1 ratio to receive either: 1) BetaBionics iLet HCL system; 2) Insulet OP 5 HCL system; 3) Tandem Control IQ HCL system, or 4) Continued MDI. All trial participants will use CGM, Block randomization, within strata defined by A1c (> vs ≤ 9%), using blocks of sizes 4 and 6, randomly permuted will be done. The groups are expected to have >20% participants screening A1c >9%.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Multiple daily injections (Active Comparator): Participants randomized into this arm will use multiple daily injections of insulin.
  Interventions: Other: Study clinician/educator visit
- BetaBionics iLet HCL system (Experimental): Participants randomized into this arm will use the BetaBionics iLet HCL system.
  Interventions: Device: Device specific training
- Insulet OP 5 HCL system (Experimental): Participants randomized into this arm will use the Insulet OP 5 HCL system.
  Interventions: Device: Device specific training
- Tandem Control IQ HCL system (Experimental): Participants randomized into this arm will use the Tandem Control IQ HCL system.
  Interventions: Device: Device specific training

INTERVENTIONS:
Device: Device specific training — Device-specific training materials from the manufactures will be used. The study clinician/pump trainer will use a pump readiness check-list to evaluate the training needs.
  Arms: BetaBionics iLet HCL system; Insulet OP 5 HCL system; Tandem Control IQ HCL system
Other: Study clinician/educator visit — Participants will receive insulin dose and other diabetes management guidance.
  Arms: Multiple daily injections

SUMMARY:
Minoritized individuals with type 1 diabetes (T1D) have approximately 2% higher average A1c levels and twice the rate of hospitalizations, complications, and mortality as their white counterparts. However, the efficacy trials establishing the benefits of hybrid closed loop (HCL) pump therapy in T1D have been in more socially advantaged and predominantly non-Hispanic white patients. Use of this technology by individuals with T1D from underserved communities remains very low.

The investigators plan to conduct a randomized effectiveness trial - with broader eligibility criteria (including markedly elevated A1c) and longer follow up than the previous HCL efficacy trials - to evaluate the benefits, safety risks and treatment complications of HCL use in underserved adults with T1D. A comprehensive mixed-methods approach will be implemented to capture information about the user experience.

Participants will be randomized (3:1 ratio) to one of three FDA-approved HCL systems or continuous glucose monitoring and multiple daily injection therapy. Subjects will be followed for 9 months to collect data on effectiveness (glucose % time-in-range 70-180 mg/dL and % time < 70 mg/dL), safety (diabetic ketoacidosis and severe hypoglycemia events) and patient experience using the systems (including benefits and burdens, the impact of life stressors on HCL use, and how the match between HCL system functionality and the individual's needs and expectations impacts on user experience).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T1D for at least 12 months, on MDI for at least 6 months;
* A1c >7.5% with no upper limit at screening (The investigator will consider the participant A1c level, compliance with current diabetes management, and prior acute diabetic complications. For this reason, there is no upper limit on A1c specified for eligibility);
* Able to understand, speak and read English (Given the language limitations in currently available pump interfaces, subjects who are not able to understand written English will not be eligible);
* Willingness to use either lispro or aspart insulin and no other insulin or new non-insulin diabetes pharmacotherapy during the study;
* Total daily dose of insulin of at least 10 units/day;
* Investigator believes that the participant will be able to successfully adhere to the study protocol.

Exclusion Criteria:

* Current use of insulin pump or closed loop insulin pump system;
* Unable to provide informed consent;
* Currently taking hydroxyurea or have medical condition that may necessitate use of hydroxyurea;
* Current use of SGLT-2 inhibitors or sulfonylureas (If using GLP-1RA, pramlintide or metformin, must be on a stable dose for 3 months prior to enrollment);
* Tape allergy or skin condition precluding use of pump or CGM;
* Females who are pregnant or intending to become pregnant (since automated algorithm adaption for some of the HCL systems used in the trial cannot be configured to adjust to changing insulin demands of pregnancy);
* Current renal dialysis or plan to begin renal dialysis during study. Most recent eGFR <30 ml/min is exclusionary (within last 2 years is acceptable);
* Active cancer treatment;
* Extreme visual or hearing impairment that would impair ability to use CGM and pump;
* Cognitive concerns;
* Significant psychiatric diagnosis or substance abuse disorder that in the investigator's opinion impairs ability of the individual to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Glucose time-in-range (TIR) of 70-180 mg/dL | baseline, 39 weeks
  The glucose TIR will be measured over 2 weeks using continuous glucose monitoring (CGM).

SECONDARY OUTCOMES:
Glucose time < 70 mg/dL | baseline, 39 weeks
  The glucose time <70 mg/dL will be measured over 2 weeks using continuous glucose monitoring (CGM).
Glucose management indicator (GMI) | baseline, 39 weeks
  The GMI will be measured using continuous glucose monitoring (CGM).
A1C | baseline, 39 weeks
  A hemoglobin A1C test is a blood test that measures a person's average blood glucose level over the previous three months.
Body weight | baseline, 39 weeks
  Participants' body weight will be measured and recorded.
Diabetic Ketoacidosis events | baseline, 39 weeks
  Events of diabetic ketoacidosis with be abstracted electronic and medical record review and from patient report.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wolpert, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No